CLINICAL TRIAL: NCT06590181
Title: Comparing the Effects of Yoga Nidra to Yoga Nidra With Pain Acceptance Intention and Motor Imagery on Pain Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, Abigail Wilson, Assistant Professor, University of Central Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YN10
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Chronic Pain
Keywords: chronic pain; meditation
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yoga Nidra (Experimental): This protocol is derived from The Origin and Clinical Relevance of Yoga Nidra (Pandi-Perumal, S. R. 2022) and is approximately 20 minutes total time.
  Interventions: Other: Yoga Nidra
- Yoga Nidra and Pain Acceptance Intention (Active Comparator): Yoga Nidra plus a Pain Acceptance Intention.
  Interventions: Other: Yoga Nidra with Pain Acceptance Intention
- Yoga Nidra with Pain Acceptance Intervention and Motor Imagery (Active Comparator): Yoga Nidra plus pain acceptance and motor imagery
  Interventions: Other: Yoga Nidra with Pain Acceptance Intervention and Motor Imagery

INTERVENTIONS:
Other: Yoga Nidra — This protocol is derived from The Origin and Clinical Relevance of Yoga Nidra (Pandi-Perumal, S. R. 2022)
  Arms: Yoga Nidra
Other: Yoga Nidra with Pain Acceptance Intention — Yoga Nidra with Pain Acceptance Intention
  Arms: Yoga Nidra and Pain Acceptance Intention
Other: Yoga Nidra with Pain Acceptance Intervention and Motor Imagery — Yoga Nidra with Pain Acceptance Intervention and Motor Imagery
  Arms: Yoga Nidra with Pain Acceptance Intervention and Motor Imagery

SUMMARY:
Yoga Nidra is a scripted mind-body intervention (MBI) that uses guided relaxation technique in a reproducible sequence of mechanisms that naturally produce a parasympathetic response. This is a randomized controlled trial in which participants will be randomly assigned to one of three interventions: 1) yoga nidra (Yoga Nidra Script Basic), 2) yoga nidra with pain acceptance (Yoga Nidra Acceptance Intention), 3) yoga nidra with pain acceptance and Explicit Motor Imagery (Yoga Nidra Acceptance Intention and Visualization).

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain in the neck, low back, shoulder, hip, elbow, knee, wrist, or ankle that has lasted for over three months
* Pain intensity rated as 3/10 or higher in the past 24 hours (0=no pain, 10=worst pain imaginable)

Exclusion Criteria:

* non-English speaking
* systemic medical conditions that affect sensation (such as uncontrolled diabetes)
* History of surgery or fracture within the past six months
* any blood clotting disorders (such as hemophilia)
* any contraindication to the application of ice (blood pressure > 140/90 mmHg, cold urticaria, cryoglobulinemia, paroxysmal cold hemoglobinuria, circulatory compromise)
* Exceed pressure and heat sensory thresholds
* Unable to access internet or email
* Pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Pressure Pain Threshold | Pre/Post intervention, Day 1
  A computerized pressure algometer (AlgoMed, Ramat Yishai, Israel) with a 1 cm diameter rubber tip will be applied to the upper trapezius.
Temporal Summation | Pre/Post intervention, Day 1
  Change in pain ratings during 10 heat pulses will be recorded.
Conditioned Pain Modulation | Pre/Post intervention, Day 1
  Pressure pain threshold after a cold water immersion task.
Heat Pain Threshold | Pre/Post intervention, Day 1
  Participants will report when comfortable heat becomes painful by pressing a button. Temperature in degrees Celsius will be recorded at threshold

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Anderson, PT, DPT, PhD, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No